CLINICAL TRIAL: NCT00615498
Title: Study to Evaluate the Effects of Weight Loss on Airway Inflammation and Mechanics in Subjects With Asthma
Brief Title: Study to Evaluate the Effects of Weight Loss on Airway Inflammation and Mechanics in Subjects With Asthma (Asthma-Bariatric Surgery Study)
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Fernando Holguin, MD, MPH, Emory University
Other Study IDs: IRB00000064
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: Asthma, obesity, bariatric
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and exhaled breath condensate samples will obtained at all time points (baseline, 1 month, 6 months, and 1 year.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical cases: Subjects who are undergoing bariatric surgery
- Controls: Subjects who qualify for bariatric surgery but do not undergo the procedure

SUMMARY:
Current research shows that obesity greatly increases the risk of developing asthma. Although the two conditions are clearly related, experts do not fully understand why they are linked. Some researchers believe that hormones released in the fat cells (adipokines) play a role. Others believe that excess weight pressing on the lungs triggers the hyperreactive response in the airways that is typical of asthma.

The goal of the Asthma-Bariatric Surgery Study is to determine how weight loss affects lung function and various biological parameters. Bariatric (weight loss) surgery refers to the various surgical procedures performed to treat obesity. Specifically, this study is designed to answer the following questions:

* Does bariatric surgery help patients control their asthma?
* How much asthma control can be achieved through weight loss?
* How does weight loss influence lung function?

Participants in this observational research study will be asked to complete study visits at enrollment, 1 month, 6 months, and 12 months. Questionnaires, pulmonary function tests, and blood samples will be required at each time point.

This research study is observational only; it does not cover the cost of (or provide) bariatric surgery. Optional genetic and bronchoscopy substudies are included as well.

DETAILED DESCRIPTION:
This study is designed to explain the unexpected effects of obesity on NO bioavailability in the airways of asthmatics: Specifically, that obesity induces systemic oxidative stress in part through increased production of reactive oxygen species (ROS) in adipose tissue and, in parallel (or as a consequence), increased systemic levels of tumor necrosis factor (TNF-α)and 8-isoprostanes. Furthermore, it creates an imbalance in the regulation of protective anti-oxidant thiol/disulfide pairs such as glutathione/glutathione disulfide. We hypothesize that in asthmatics, the lung is a target-organ of this obesity-related systemic oxidative stress. This is manifested as increased oxidation of airway NO into nitrate and reactive nitrogen species (RNS) including peroxynitrate and nitrotyrosine, thereby reducing NO bioavailability and exhaled NO levels. NO has many key physiological properties including bronchodilation, anti-tumoral/bactericidal activity, and anti-inflammatory and anti-oxidative activity. Thus, reduced NO bioavailability in obese asthmatics could favor increased bronchoconstriction and impair the lung's ability to respond to further oxidative or inflammatory challenges. Therefore, we hypothesize that: 1) obesity causes redox stress in the airway, which in turn decreases the bioavailability of NO by shunting it into RNS, 2) that weight loss will decrease systemic oxidative stress and thereby increase NO bioavailability due to decreased oxidation into RNS, and 3) that by decreasing systemic oxidative stress, weight loss will reduce bronchial hyper-reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, or a limited smoking history
* Meet criteria for bariatric surgery according to NIH guidelines

Exclusion Criteria:

* Illicit drug use
* Greater than 10 pack-year history of cigarette smoking
* Other significant lung pathology
* Other significant non-pulmonary co-morbidities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese asthmatics
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To measure levels of exhaled nitric oxide, reactive nitrogen species, exhaled biomarkers of lipid peroxidation, asthma quality of life, airway function (spirometry and response to methacholine), and degree of asthma control | Enrollment, 1 month, 6 months, and 1 year
To measure systemic markers of redox stress and inflammation, including plasma levels of adipokines, adiposity-related cytokines (IL-6, TNF-α), GSH/GSSG, 8-isoprostanes, and leukotrienes | Enrollment, 1 month, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Emory Crawford Long Hospital, Clinical Research Center, Atlanta, Georgia, United States